CLINICAL TRIAL: NCT04362046
Title: Fertility Preservation Using Endomyometrial Resection for Atypical Hyperplasia and Low Grade, Stage 1A, Endometrial Cancer
Brief Title: Fertility Sparing Management of EndomeTrial Cancer and Hyperplasia
Acronym: FETCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vancouver Coastal Health Research Institute (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Mark Carey, Clinical Professor, Vancouver Coastal Health Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H17-00780
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Endometrial Hyperplasia; Endometrial Cancer; Gynecologic Cancer
Keywords: Fertility preservation; Hysteroscopic uterine resection; High-dose progesterone
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hysteroscopic uterine resection (Experimental): This is a prospective single-arm surgical intervention trial.
  Interventions: Procedure: Hysteroscopic uterine resection

INTERVENTIONS:
Procedure: Hysteroscopic uterine resection — Hysteroscopic Resection will be evaluated as a fertility-sparing treatment for patients with early Endometrial Cancer or Endometrial Hyperplasia (atypical or persisting typical) who fail progestin therapy. Failure of progesterone therapy is defined as: (a) Unsuccessful eradication of hyperplasia or cancer in the uterus or (b) Intolerance to the side effects of th hormone therapy.
  HR is a common gynecologic procedure that is offered to women for treatment of several benign gynecologic conditions. The conduct, risks, and complications of it are well-understood. In relation to this protocol, it is the indication for HR that constitutes the experimental intervention including the assessment of it's outcome. Patients deemed appropriate for hysteroscopic endomyometrial resection will be counselled on the nature of the procedure along with its risks and complications.

SUMMARY:
This study protocol evaluates the use of hysteroscopic endomyometrial resection in women diagnosed with atypical endometrial hyperplasia or grade I endometrial cancer who have not responded to anti-hormone therapy. Patients in this study wish to preserve fertility.

DETAILED DESCRIPTION:
Endometrial cancer (EC) is the most common gynecological cancer among Canadian women. This cancer often arises from a precursor lesion called atypical endometrial hyperplasia (AH). Hysterectomy is the most effective treatment for EC and AH. It is well recognized that EC may be diagnosed in younger women of child-bearing age. The diagnosis of EC or AH in these younger women is devastating as a hysterectomy is frequently required. Though some of these women respond to high-dose progestin treatment, the failure rate is high (60%), necessitating surgery. Recent case series show that some women with AH and early EC can be treated by resecting the precursor lesion of the early cancerous area in the uterus by hysteroscopy without the need for hysterectomy. The fertility-sparing approach is outlined in this research protocol.This is a multidisciplinary research project with input from gynaecologic oncology, general gynaecology, reproductive endocrinology and infertility, and pathology. Our hypothesis is that hysteroscopic resection (HR) is a safe and effective treatment for AH or EC in women who want to preserve their fertility and have not been successfully treated using progestin therapy. Patients will be closely monitored to ensure that this is a safe and effective treatment option.

ELIGIBILITY:
All candidates for this protocol must have an adequate trial of anti-hormone therapy prior to hysteroscopic resection. In cases of EC, the minimum trial is 6 months of high-dose progestin. In cases of AH, being that this is a benign condition (pre-malignant), patients may not require a full 6 months of anti-hormone therapy. All patients must have a pre-HR hysteroscopic evaluation to confirm that they are suitable candidates for this study. Patients being considered for the experimental intervention (hysteroscopic resection) will be reviewed and discussed by the study committee in order to ensure that the following criterion are met in order to proceed with the surgical resection:

Inclusion criteria:

* Age less than 40 years
* Pathologist confirmed biopsy evidence of one of the following:

  1. Grade I endometrial endometrioid adrenocarcinoma (EC) with less than 1/3 of the endometrial surface involved.
  2. Atypical endometrial hyperplasia (AH)
* MRI demonstrating less than 1/3 myometrial invasion if the patient has EC
* Absence of significant surgical co-morbidities e.g. pulmonary hypertension, significant cardiac valvular disease, or contraindication to surgery.
* Desire to preserve fertility
* Reasonable chance to conceive based on consultation with an infertility specialist
* Adequate dose and duration of progesterone therapy prior to enrolment:
* Adequate dose:

  1. Medroxyprogesterone acetate (Provera; 200mg/day)
  2. Megestrol acetate (Megace; 160mg/day)
* Adequate duration: 6 months
* Failure of progestin therapy defined as:

  1. Unsuccessful eradication of hyperplasia or cancer in the uterus
  2. Intolerance to the side effects
* Signed informed consent

Exclusion criteria:

* Age 40 years and over
* Grade 2 or 3 endometrioid endometrial adenocarcinoma or non-endometrioid pathology
* Greater than 1/3 involvement of the endometrial surface in patients with Grade I EC
* Women who are not able to provide informed consent
* Women without pathologic confirmation of low-grade endometrioid carcinoma or AH
* Myometrial invasion on MRI greater than 1/3 total myometrial thickness.
* MRI evidence of ovarian or adnexal involvement
* The diagnosis of another cancer or medical condition that would interfere with the assessment of the hysteroscopic surgery success rates.
* Significant underlying fertility impairment that would significantly interfere with the success rate of HR

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study being conducted on women who have Grade 1 endometrial cancer or atypical endometrial hyperplasia
Enrollment: 30 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Conception rate of women attempting pregnancy | 3 years post-resection
  live births / women attempting pregnancy
Overall conception rate | 3 years post-resection
  live births / all women participating in study, including those who failed hysteroscopic resection and have a hysterectomy
Local disease control rate (short-term failure of hysteroscopic resection) | 3 months post-resection
  Patients with persisting atypical hyperplasia or Grade I endometrial cancer / patients treated with hysteroscopic resection
Distant disease control rate (long-term failure of hysteroscopic resection) | 3 years post-resection
  patients developing distant recurrence / patients treated with hysteroscopic resection

SECONDARY OUTCOMES:
Complications/side-effects | 3 years post-resection
  The investigators will tabulate complications/side-effects of the procedure such as the rate of uterine perforation, uterine adhesion, procedure infection, and others.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Carey, MD, Principal Investigator — Vancouver Coastal Health
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
The information in database/registry is anonymized. Inadvertent disclosure of the data poses no risk to patients.